CLINICAL TRIAL: NCT00109109
Title: Phase II Clinical Trial of Oral Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Advanced Multiple Myeloma
Brief Title: A Clinical Trial of Oral Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Advanced Multiple Myeloma (0683-004)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 0683-004; 2005_013
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Vorinostat

INTERVENTIONS:
Drug: MK0683, vorinostat, Suberoylanilide Hydroxamic Acid (SAHA) / Duration of Treatment - Up to 8 Cycles or 6 months

SUMMARY:
The purposes of this study are:

* To determine the maximum tolerated dose (MTD) of SAHA administered every 12 hours for 14 consecutive days followed by 7 days of rest during the first two cycles (i.e., first 6 weeks) in patients with advanced multiple myeloma;
* To assess the safety and overall response rate to SAHA in patients with advanced multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with refractory or relapsed multiple myeloma, ECOG performance status 0-2 (ECOG)
* Adequate bone marrow reserve
* Adequate hepatic and renal function
* Ability to swallow capsules
* 3 weeks or more from prior chemotherapy and have recovered from prior toxicities

Exclusion Criteria:

* Patients who plan to go for bone marrow transplant within 4 weeks of start of treatment
* Patients with prior treatment with other investigational agents with a similar anti-tumor mechanism
* Patients with other active/uncontrolled clinically significant illnesses
* Pregnant or nursing female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-12-01 (Actual); Primary Completion 2006-02-14 (Actual); Study Completion 2006-02-14 (Actual)

PRIMARY OUTCOMES:
PHASE I: Maximum tolerated dose (MTD) of vorinostat in patients with advanced multiple myeloma.
PHASE II: Safety and overall response rate to SAHA in patients with advanced multiple myeloma.

SECONDARY OUTCOMES:
1) Anti-tumor activity in patients with advanced multiple myeloma; 2) Biological effects of SAHA in peripheral mononuclear cells and bone marrow plasma cells; 3) Correlation of biological effects of SAHA with serum drug concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Richardson P, Mitsiades C, Colson K, Reilly E, McBride L, Chiao J, Sun L, Ricker J, Rizvi S, Oerth C, Atkins B, Fearen I, Anderson K, Siegel D. Phase I trial of oral vorinostat (suberoylanilide hydroxamic acid, SAHA) in patients with advanced multiple myeloma. Leuk Lymphoma. 2008 Mar;49(3):502-7. doi: 10.1080/10428190701817258. PMID 18297527
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/policies-perspectives.html